CLINICAL TRIAL: NCT03632408
Title: The Effect of Alcohol Hangover and Night-time Zopiclone on Next-morning Spatial Perception in Healthy Young Volunteers
Brief Title: Hangover and Residual Zopiclone Effect on Spatial Perception
Acronym: SEKO-A
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Petri Vainio (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor-Investigator, Petri Vainio, Assistant professor, Turku University Hospital
Organization: Turku University Hospital (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: T271
Record Dates: First submitted 2018-08-07; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Healthy; Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — zopiclone; hang protein, Drosophila

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Alcohol not masked Zopiclone and placebo capsulated, identical in weight and appearance Third party generated code only available to pharmacy and in case of emergency
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Zopiclone — Oral, single dose, 7.5 mg
Behavioral: hangover — as per subjects choice to consume alcohol
Drug: Placebo oral capsule — oral

SUMMARY:
Hangover after recreational alcohol use, residual effect of zopiclone and placebo compared in terms of spatial perception, psychomotor tests and simulated driving ability. Three recording visits plus screening included.

ELIGIBILITY:
Inclusion Criteria:

* weight >45 kg
* likely to experience and predict alcohol hangover within the next five weeks
* no childbearing potential of negative pregnancy test at screening
* a valid driving license

Exclusion Criteria:

* breastfeeding
* infection with HCV, HBV or HIV
* a medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation
* suspected or current drug or alcohol abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Driving error rate | Day 1
  Driving error rate
Number of erroneous responses to peripheral visual stimuli during driving | Day 1
  Number of erroneous responses to peripheral visual stimuli during driving

SECONDARY OUTCOMES:
digit symbol substitution | Day 1
  digit symbol substitution test
drug concentration | Day 1
  concentration of zopiclone in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Petri J Vainio, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Teutori clinical trial facility, Turku, Finland